CLINICAL TRIAL: NCT02619942
Title: A Multicenter, Prospective, Randomized Clinical Trial to Investigate the Radical Extent of Lymphadenectomy: D2 Dissection vs. Complete Mesocolic Excision, of LAparoscopic Right Colectomy for Right-sided Colon Cancer.
Brief Title: Investigate the Radical Extent of Lymphadenectomy of LAparoscopic Right Colectomy for Colon Cancer(RELARC).
Acronym: RELARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University Cancer Hospital & Institute (Other); Beijing Friendship Hospital (Other); Xuanwu Hospital, Beijing (Other); Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Hospital of Jilin University (Other); Nanfang Hospital, Southern Medical University (Other); Fujian Medical University Union Hospital (Other); Peking Union Medical College (Other); Peking University People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); RenJi Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, XIAO Yi, MD, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RELARC
Record Dates: First submitted 2015-11-29; First posted 2015-12-02 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer
Keywords: Right colon cancer, Survival, Laparoscopic surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 radical operation group (Active Comparator): In D2 radical operation group(D2), the mesocolon should be removed and the dissection involves the paracolon and intermediate lymph nodes, which along the feeding vessels.
  Interventions: Procedure: D2 radical operation
- CME group (Experimental): In complete mesocolic excision group (CME), in addition to D2 dissection, the whole mesocolon, from ascending colon to right half transverse colon, as well as the central lymph nodesmshould be entirely removed.
  Interventions: Procedure: Complete mesocolic excision (CME)

INTERVENTIONS:
Procedure: D2 radical operation — In D2 radical operation group(D2), the lymph node dissection is based on ligating the supplying vessels close to the right-side of superior mesenteric vein and clean up the surrounding lymph node and adipose tissue.
  Arms: D2 radical operation group
Procedure: Complete mesocolic excision (CME) — In complete mesocolic excision group (CME), the dissecting extent includes the lymphatic and fat tissues surrounding the root of ascending mesocolon, which situated on the surface of superior mesenteric vein, and the root of right half of transverse mesocolon, which situated on the surface of pancreas neck.
  Arms: CME group

SUMMARY:
To investigate whether extended lymphadenectomy (CME) in laparoscopic colectomy could improve disease-free survival in patients with right colon cancer, compared with standard D2 radical operation.

DETAILED DESCRIPTION:
Our study design is a two-arm, parallel-group, single-blind randomized clinical trial. The enrolled colon cancer patients would be divided into the intervention group (CME group) and control group (D2 radical operation group).

The postoperative adjuvant chemotherapy is determined by the pathological results. For patients of stage Ⅲ and patients of stage Ⅱ with unfavorable histologic features, six months of adjuvant chemotherapy of XELOX or fluorouracil-based regimen are recommended.

The postoperative examination should be performed every four months in the first two years and every six months in the following three years, to exclude local recurrence and distant metastasis.

Our study is expected to last five years, of which two years for recruiting patients, three years for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suitable for curative surgery 18-75years old
2. ASA grade I-III
3. Qualitative diagnosis: a pathological diagnosis of adenocarcinoma;
4. Localization diagnosis: the tumor located between the cecum and the right 1/3 of transverse colon;
5. Enhanced CT scan of chest, abdominal and pelvic cavity: assessment of tumor stage is T2-T4N0 or TanyN+; there is no distant metastasis.
6. Informed consent

Exclusion Criteria:

1. Simultaneous or simultaneous multiple primary colorectal cancer;
2. Preoperative imaging examination results show: (1) colon cancer of stage T1N0; (2) enlargement of lymph node at the root of mesocolon, in which case the D3 radical operation must be performed;
3. Preoperative imaging examination results show: (1) Tumor involves the surrounding organs and combined organ resection need to be done; (2)distant metastasis; (3)unable to perform R0 resection;
4. History of any other malignant tumor in recent 5 years, except for cervical carcinoma in situ which has been cured, basal cell carcinoma or squamous cell carcinoma of skin;
5. Patients need emergency operation;
6. Not suitable for laparoscopic surgery (i.e., extensive adhesion caused by abdominal surgery, not suitable for artificial pneumoperitoneum, etc).
7. Informed consent refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Estimated)
Dates: Start 2016-01-09 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2022-12-26 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years
  The proportion of patients with no disease recurrence and metastasis after 3 years of surgery

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Complications occurring within 30 days after surgery
Postoperative mortality | 30 days
  Death occurred within 30 days after surgery
3 years overall survival | 3 years
  The proportion of patients who survived 3 years after surgery
Metastasis rate of central lymph node (3rd station) | 7 days
  Metastasis rate of central lymph node (3rd station)

CONTACTS AND LOCATIONS:
Overall Officials: Yi XIAO, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lai XU, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li K, Li H, Wu A, Zang L, Zhang G, Xu L, Lu J, Xing J, Feng B, Sun Y, Du X, Chi P, Xu J, Wang Z, Zhang Y, Zhang Z, Zheng M, Su X, Xiao Y; RELARC Study Group. Long-Term Survival on Extent of Lymphadenectomy for Right-Sided Colon Cancer: Five-Year Follow-up Results of a Randomized Controlled Trial (RELARC Trial). Ann Surg. 2025 Sep 12. doi: 10.1097/SLA.0000000000006941. Online ahead of print. PMID 40938728
- [Derived] Lu J, Xing J, Zang L, Zhang C, Xu L, Zhang G, He Z, Sun Y, Feng Y, Du X, Hu S, Chi P, Huang Y, Wang Z, Zhong M, Wu A, Zhu A, Li F, Xu J, Kang L, Suo J, Deng H, Ye Y, Ding K, Xu T, Zhang Y, Zhang Z, Zheng M, Su X, Xiao Y; RELARC study group. Extent of Lymphadenectomy for Surgical Management of Right-Sided Colon Cancer: The Randomized Phase III RELARC Trial. J Clin Oncol. 2024 Nov 20;42(33):3957-3966. doi: 10.1200/JCO.24.00393. Epub 2024 Aug 27. PMID 39190853
- [Derived] Sun Z, Zhang G, Lu J, Wu B, Lin G, Xiao Y, Xu L. Risk Factors for Postoperative Complications of Laparoscopic Right Colectomy: A Post Hoc Analysis of the RELARC Trial. Dis Colon Rectum. 2024 Sep 1;67(9):1194-1200. doi: 10.1097/DCR.0000000000003331. Epub 2024 May 21. PMID 38773832
- [Derived] Xu L, Su X, He Z, Zhang C, Lu J, Zhang G, Sun Y, Du X, Chi P, Wang Z, Zhong M, Wu A, Zhu A, Li F, Xu J, Kang L, Suo J, Deng H, Ye Y, Ding K, Xu T, Zhang Z, Zheng M, Xiao Y; RELARC Study Group. Short-term outcomes of complete mesocolic excision versus D2 dissection in patients undergoing laparoscopic colectomy for right colon cancer (RELARC): a randomised, controlled, phase 3, superiority trial. Lancet Oncol. 2021 Mar;22(3):391-401. doi: 10.1016/S1470-2045(20)30685-9. Epub 2021 Feb 12. PMID 33587893
- [Derived] Lu JY, Xu L, Xue HD, Zhou WX, Xu T, Qiu HZ, Wu B, Lin GL, Xiao Y. The Radical Extent of lymphadenectomy - D2 dissection versus complete mesocolic excision of LAparoscopic Right Colectomy for right-sided colon cancer (RELARC) trial: study protocol for a randomized controlled trial. Trials. 2016 Dec 8;17(1):582. doi: 10.1186/s13063-016-1710-9. PMID 27931247
- See also: The Radical Extent of lymphadenectomy D2 dissection versus complete mesocolic excision of LAparoscopic Right Colectomy for right-sided colon cancer (RELARC) trial: study protocol for a randomized controlled tria — http://www.trialsjournal.com/content/17/1/582
- Available data/document: Study Protocol — http://www.trialsjournal.com/content/17/1/582